CLINICAL TRIAL: NCT06115915
Title: AIVertigo: Automated Differential Diagnosis of Vertigo Using Video-oculography and Advanced Artificial Intelligence-based Triage
Brief Title: AIVertigo: AIVertigo: Automated Differential Diagnosis of Vertigo Using Video-oculography and Advanced Artificial Intelligence-based Triage
Status: Completed | Type: Observational
Sponsor: Neurobit Technologies Co., Ltd. (Industry)
Collaborators: Taipei Medical University (Other); Buddhist Tzu Chi Medical Foundation (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2020061901SAMD
Record Dates: First submitted 2023-10-28; First posted 2023-11-03 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-11

CONDITIONS: Vertigo
Keywords: Vertigo; Videonystagmography (VNG); Software as Medical Device (SaMD); Computer-Aided Triage and Notification (CADt); Artificial Intelligence/Machine Learning (AI/ML)
MeSH Terms: conditions — Vertigo

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The eye movement records and vestibular pulse examinations obtained from patients with dizziness can provide characteristic parameters and features of eye movements and vestibular reflexes. These can assist specialized physicians in diagnosing various forms of dizziness disorders. Through extensive analysis of databases, a disease prediction model can be established, significantly lowering the diagnostic barriers for non-specialist doctors, thereby enabling their diagnostic capabilities to approach that of experts.

DETAILED DESCRIPTION:
Investigators analyze the VOG and vHIT data of vertigo patients in the dizziness clinics of two medical institutions: Shuang Ho Hospital (SHH) between June 2020 and June 2021 and Taichung Tzu Chi Hospital (TTCH) between July 2019 and August 2020, respectively. The institutional review boards of SHH (TMU-JIRB No. N202005118) and TTCH (REC 109-64) approved the study. All patients received structuralized history taking, neurological examinations, neuro-otological examinations, VOG and vHIT. All patients who had focal neurological symptoms/signs or central vestibular/oculomotor signs underwent brain MRI. Final diagnoses were conducted after the comprehensive studies above. The patients who did not finish VOG tests or vHIT or who had invalid data in VOG or vHIT, as well as those with uncertain final diagnoses, were excluded from the study.

According to the final diagnoses, all patients were further classified into "benign vertigo" and "dangerous vertigo" groups as the reference standard of this study. Benign vertigo is defined as vertigo that is not caused by any serious underlying condition and is generally considered harmless or self-limiting. It includes all peripheral-type vertigo and "benign" central-type vertigo without structural lesions in the brain, such as vestibular migraine and persistent postural-perceptual dizziness. However, dangerous vertigo is defined as the vertigo that is caused by a potentially severe or life-threatening underlying condition that requires immediate medical attention and intervention. It includes central-type vertigo with compatible structural lesions in the brain MRI, vertebrobasilar insufficiency with compatible stenotic arteries in MRI, and cerebellar degeneration with brain atrophy in MRI or apparent cerebellar ataxia. The classification of benign or dangerous vertigo was performed by two neurologists with expertise in dizziness and vertigo at each medical institution (SHH and TTCH) after they reviewed the clinical information and final diagnoses. In case they had differing opinions, they reached a consensus via video conferences. Otherwise, the clinical workflow was in accordance with the standard procedures of each medical institution.

ELIGIBILITY:
Inclusion Criteria:

* Dizziness receiving medical treatment at the Neurology and Otolaryngology departments' outpatient clinics including cases transferred from the emergency department to outpatient clinics.
* Inpatient wards (including cases transferred from the emergency department to hospitalization) of the Neurology and Otolaryngology departments.

Exclusion Criteria:

* With prosthetic eyes.
* Uncorrected visual acuity below 0.1.
* Severe hearing or cognitive impairments preventing examination.
* Severe cervical spine conditions precluding examination.
* Unable to sit for prolonged periods.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients with dizziness who seek treatment at the Neurology or Otolaryngology outpatient clinics or are admitted to Shuang Ho Hospital are potential candidates for enrollment. Patients who meet the inclusion criteria and have the research purpose and process explained by a physician or research assistant, agree to participate in this study, and complete the informed consent form will be considered eligible for enrollment.
Sampling Method: Probability Sample
Enrollment: 391 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-06-18 (Actual); Study Completion 2021-06-18 (Actual)

PRIMARY OUTCOMES:
Performance Indices | 2 hour per individual
  1. Sensitivity, specificity, positive predictive value, and negative predictive value of combined parameters of eye movement and vestibular reflex in screening various types of vestibular disorders.
  2. Sensitivity, specificity, positive predictive value, and negative predictive value of combined parameters of eye movement and vestibular reflex in screening various types of vestibular disorders cross different medical institution

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Medical University-Shuang Ho Hospital,Ministry of Health and Welfare, New Taipei City, Taiwan